CLINICAL TRIAL: NCT04852406
Title: Effect of Protocol-based Management on Perioperative Outcomes in Patients With Chronic Antithrombotic Therapy: a Pragmatic Interventional Study
Brief Title: Protocol-based Management and Perioperative Outcomes in Patients With Chronic Antithrombotic Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-432
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Antithrombotic Therapy; Perioperative Care; Perioperative Outcomes
Keywords: perioperative care; antithrombotic therapy; perioperative outcomes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this group receive protocol-based management of perioperative antithrombotic therapy.
  Interventions: Drug: Protocol-based management of perioperative antithrombotic therapy
- Control group (Sham Comparator): Participants in this group receive routine management of perioperative antithrombotic therapy.
  Interventions: Drug: Routine management of perioperative antithrombotic therapy

INTERVENTIONS:
Drug: Protocol-based management of perioperative antithrombotic therapy — Perioperative antithrombotic therapy is managed according to the latest expert consensus published in the Chinese Medical Journal, 2020.
  Other Names: Protocol-based management
  Arms: Intervention group
Drug: Routine management of perioperative antithrombotic therapy — Perioperative antithrombotic therapy is managed according to current routine practice.
  Other Names: Routine management
  Arms: Control group

SUMMARY:
The purpose of this pragmatic interventional study is to evaluate whether a protocol-based management of antithrombotic drugs can reduce a composite of perioperative outcomes in patients with chronic antithrombotic therapy before surgery.

DETAILED DESCRIPTION:
Aging population and chronic medical disease make the management of surgical patients more complex. About one tenth of patients scheduled for surgery are taking antithrombotic medications. Coagulation disturbance induced by these medications may increase the risk of bleeding, whereas withholding these medications may increase the risk of thrombotic events. It is a dilemma when managing these patients.

The guidelines and expert consensus published by multiple disciplinary teams constitute the perioperative antithrombotic management protocols. However, the effects of perioperative antithrombotic management guided by these guidelines or expert consensus are seldom reported. The investigators hypothesize that a protocol-based perioperative antithrombotic management can benefit patients with chronic antithrombotic therapy before surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with continuing antithrombotic therapy (including antiplatelet and/or anticoagulant therapies) for cardiovascular and cerebrovascular diseases for more than 2 weeks.
* 2. Patients who have one or more of the following situations: (1) non-valvular atrial fibrillation with a CHA2DS2-VASc score >4; (2) post-artificial valve replacement (including mitral valve, ball-cage valve or tilting disc aortic valve); (3) venous thromboembolism occurred within 1 year, or venous thromboembolism with other high-risk factors which require long-term anticoagulation treatment; (4) coronary heart disease with coronary stent implantation, thrombolytic therapy or other coronary procedures within 2 years, or who had undergone coronary artery bypass grafting within 1 year, or who experienced myocardial infarction or acute coronary syndrome within 1 year; (5) a history of stroke/transient ischemic accident within 1 year, or a history of cervical or intracranial revascularization treatment within 1 year; (6) peripheral arterial disease.
* 3. Patients who are scheduled to undergo intra-abdominal surgery (including general and urologic surgery).
* 4. Patients who sign written informed consents.

Exclusion Criteria:

* 1. Refuse to participate.
* 2. Emergency surgery.
* 3. Unable to complete the preoperative assessment and follow-up plan.
* 4. Other reasons that are considered unsuitable for study participation by the investigators or the attending doctors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 526 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of a composite outcome including major bleeding and major adverse cardiovascular or cerebrovascular events | Up to 30 days after surgery
  Major bleeding indicates bleeding of type 2 or higher on the BARC (Bleeding Academic Research Consortium) criteria. Major adverse cardiovascular or cerebrovascular events indicate acute coronary syndrome, acute myocardium infarction, ischemic stroke/transient ischemic attack, systemic arterial embolism, pulmonary embolism, or all-cause death.

SECONDARY OUTCOMES:
Incidence of other postoperative complications | Up to 30 days after surgery
  Other postoperative complications indicate any newly occurred medical events that are harmful to patients' recovery and required therapeutic intervention, except major bleeding and major adverse cardiovascular or cerebrovascular events.
The length of hospital stay | Up to 30 days after surgery
  The length of hospital stay from admission to discharge
Total expenses during hospitalization | Up to 30 days after surgery
  Total expenses during hospitalization
All-cause mortality rate within 30 days after surgery | Up to 30 days after surgery
  All-cause mortality rate within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
on demands.

REFERENCES:
- [Background] Hornor MA, Duane TM, Ehlers AP, Jensen EH, Brown PS Jr, Pohl D, da Costa PM, Ko CY, Laronga C. American College of Surgeons' Guidelines for the Perioperative Management of Antithrombotic Medication. J Am Coll Surg. 2018 Nov;227(5):521-536.e1. doi: 10.1016/j.jamcollsurg.2018.08.183. Epub 2018 Aug 24. No abstract available. PMID 30145286
- [Background] Dubois V, Dincq AS, Douxfils J, Ickx B, Samama CM, Dogne JM, Gourdin M, Chatelain B, Mullier F, Lessire S. Perioperative management of patients on direct oral anticoagulants. Thromb J. 2017 May 15;15:14. doi: 10.1186/s12959-017-0137-1. eCollection 2017. PMID 28515674
- [Background] Torn M, Rosendaal FR. Oral anticoagulation in surgical procedures: risks and recommendations. Br J Haematol. 2003 Nov;123(4):676-82. doi: 10.1046/j.1365-2141.2003.04652.x. PMID 14616972
- [Background] Oltmann SC, Alhefdhi AY, Rajaei MH, Schneider DF, Sippel RS, Chen H. Antiplatelet and Anticoagulant Medications Significantly Increase the Risk of Postoperative Hematoma: Review of over 4500 Thyroid and Parathyroid Procedures. Ann Surg Oncol. 2016 Sep;23(9):2874-82. doi: 10.1245/s10434-016-5241-0. Epub 2016 May 2. PMID 27138383
- [Background] Yurttas T, Wanner PM, Filipovic M. Perioperative management of antithrombotic therapies. Curr Opin Anaesthesiol. 2017 Aug;30(4):466-473. doi: 10.1097/ACO.0000000000000481. PMID 28509773
- [Background] Yong JW, Yang LX, Ohene BE, Zhou YJ, Wang ZJ. Periprocedural heparin bridging in patients receiving oral anticoagulation: a systematic review and meta-analysis. BMC Cardiovasc Disord. 2017 Dec 13;17(1):295. doi: 10.1186/s12872-017-0719-7. PMID 29237411
- [Background] Childers CP, Maggard-Gibbons M, Ulloa JG, MacQueen IT, Miake-Lye IM, Shanman R, Mak S, Beroes JM, Shekelle PG. Perioperative management of antiplatelet therapy in patients undergoing non-cardiac surgery following coronary stent placement: a systematic review. Syst Rev. 2018 Jan 10;7(1):4. doi: 10.1186/s13643-017-0635-z. PMID 29321066
- [Background] Howell SJ, Hoeks SE, West RM, Wheatcroft SB, Hoeft A; OBTAIN Investigators of European Society of Anaesthesiology (ESA) Clinical Trial Network. Prospective observational cohort study of the association between antiplatelet therapy, bleeding and thrombosis in patients with coronary stents undergoing noncardiac surgery. Br J Anaesth. 2019 Feb;122(2):170-179. doi: 10.1016/j.bja.2018.09.029. Epub 2018 Dec 15. PMID 30686302
- [Background] Widimsky P, Motovska Z, Havluj L, Ondrakova M, Bartoska R, Bittner L, Dusek L, Dzupa V, Knot J, Krbec M, Mencl L, Pachl J, Grill R, Haninec P, Waldauf P, Gurlich R. Perioperative cardiovascular complications versus perioperative bleeding in consecutive patients with known cardiac disease undergoing non-cardiac surgery. Focus on antithrombotic medication. The PRAGUE-14 registry. Neth Heart J. 2014 Sep;22(9):372-9. doi: 10.1007/s12471-014-0575-3. PMID 25120211
- [Background] Cao D, Mehran R, Dangas G, Baber U, Sartori S, Chandiramani R, Stefanini GG, Angiolillo DJ, Capodanno D, Urban P, Morice MC, Krucoff M, Goel R, Roumeliotis A, Sweeny J, Sharma SK, Kini A. Validation of the Academic Research Consortium High Bleeding Risk Definition in Contemporary PCI Patients. J Am Coll Cardiol. 2020 Jun 2;75(21):2711-2722. doi: 10.1016/j.jacc.2020.03.070. PMID 32466887
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542